CLINICAL TRIAL: NCT07381517
Title: Correlation Between Oxygenation Indices (OI and Their Derivatives) and Oxygen Saturation Indices (OSI and Their Derivatives) During One-Lung Ventilation in Thoracic Surgery
Brief Title: Correlation of Oxygenation and Saturation Indices in One-Lung Ventilation
Acronym: OLV-INDICES
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Onur KARSLIOĞLU, Resident Physician in Anesthesiology, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: OLV-OXY-001
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: One-lung Ventilation (OLV)
Keywords: One-Lung Ventilation; Oxygenation; Oxygen Saturation Index; Driving Pressure; Mechanic Power; Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One-Lung Ventilation Cohort: Adult patients undergoing elective thoracic surgery requiring one-lung ventilation. All patients will be managed according to standard clinical practice. No intervention is assigned as part of this observational study.

SUMMARY:
One-lung ventilation is commonly used during thoracic surgery but is frequently associated with impaired oxygenation and altered respiratory mechanics. Traditional oxygenation indices require arterial blood gas analysis and do not fully reflect the mechanical stress applied to the lungs.

This prospective observational study aims to evaluate the correlation between oxygenation indices and oxygen saturation indices during one-lung ventilation in adult patients undergoing elective thoracic surgery. Modified indices incorporating driving pressure and mechanical power will also be assessed.

No intervention beyond standard clinical care will be applied. The findings of this study may help clarify the clinical utility of non-invasive oxygenation indices for intraoperative monitoring during one-lung ventilation.

DETAILED DESCRIPTION:
One-lung ventilation induces complex changes in pulmonary physiology, including increased intrapulmonary shunt and altered respiratory mechanics, which may challenge conventional approaches to intraoperative oxygenation assessment. While invasive oxygenation indices are widely used, their applicability during one-lung ventilation is limited by the need for arterial blood gas sampling and the lack of integration of mechanical ventilation-related stress.

Non-invasive oxygen saturation-based indices have been proposed as alternatives; however, data regarding their performance under the dynamic physiological conditions of one-lung ventilation remain scarce. Furthermore, emerging concepts in lung-protective ventilation emphasize the importance of driving pressure and mechanical power as determinants of ventilator-induced lung injury, yet these parameters are not incorporated into traditional oxygenation metrics.

In this prospective observational study, invasive and non-invasive oxygenation indices, including modified forms incorporating driving pressure and mechanical power, will be recorded simultaneously during one-lung ventilation in adult patients undergoing elective thoracic surgery. The relationships and agreement between these indices will be analyzed to assess their comparability across different levels of mechanical respiratory load.

No intervention beyond standard clinical care will be applied. Ventilatory settings and perioperative management will be determined solely by routine clinical practice. This study is designed to provide methodological insight into the intraoperative applicability of non-invasive oxygenation indices during one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients classified as ASA physical status I-III
* Patients scheduled for elective thoracic surgery requiring one-lung ventilation for at least 1 hour intraoperatively
* Patients in whom simultaneous arterial blood gas analysis and continuous SpO₂ monitoring can be performed
* Patients who have provided written informed consent

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients younger than 18 years of age
* Patients classified as ASA physical status IV or higher
* Patients with a history of previous thoracic surgery
* Patients with a body mass index (BMI) >40 kg/m² or <18 kg/m²
* Patients with advanced chronic lung disease (COPD stage III-IV)
* Patients with New York Heart Association (NYHA) class III-IV heart failure
* Patients undergoing surgery due to pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older with ASA physical status I-III who are scheduled for elective thoracic surgery requiring intraoperative one-lung ventilation for at least one hour. All participants undergo standard perioperative management with simultaneous arterial blood gas analysis and continuous pulse oximetry monitoring during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between oxygenation indices and oxygen saturation indices | During intraoperative one-lung ventilation
  Correlation between invasive oxygenation indices (oxygenation index and its derivatives) and non-invasive oxygen saturation indices (oxygen saturation index and its derivatives) measured during one-lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Onur KARSLIOĞLU, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Ataturk Sanatoryum Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lohmann T, Nietzschmann U, Kiess W. "Lady-like": is there a latent autoimmune diabetes in the young? Diabetes Care. 2000 Nov;23(11):1707-8. doi: 10.2337/diacare.23.11.1707. No abstract available. PMID 11092301
- [Result] Chiumello D, Carlesso E, Cadringher P, Caironi P, Valenza F, Polli F, Tallarini F, Cozzi P, Cressoni M, Colombo A, Marini JJ, Gattinoni L. Lung stress and strain during mechanical ventilation for acute respiratory distress syndrome. Am J Respir Crit Care Med. 2008 Aug 15;178(4):346-55. doi: 10.1164/rccm.200710-1589OC. Epub 2008 May 1. PMID 18451319
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- See also: Ankara Atatürk Sanatoryum Training and Research Hospital — https://sanatoryumdh.saglik.gov.tr/
- Available data/document: Informed Consent Form — https://sanatoryumdh.saglik.gov.tr/ — Individual participant data collected during this observational study will not be shared publicly. The study data will be used solely for the purposes defined in the approved study protocol (V3) and ethics committee approval. No supporting documents such as study protocol, statistical analysis plan, or case report forms will be made publicly available, as data sharing was not planned or approved in the informed consent process.